CLINICAL TRIAL: NCT00197496
Title: Body Weight Supported Treadmill Training Following Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Lora Giangregorio, Postdoctoral fellow/Affiliate Scientist, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIF-05055
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BWSTT (Experimental): Body weight supported treadmill training
  Interventions: Procedure: Body weight supported treadmill training
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Procedure: Body weight supported treadmill training — hip fracture patients walk on a treadmill with body weight support
  Other Names: treadmill training
  Arms: BWSTT

SUMMARY:
Achieving independent ambulation is an important goal of hip fracture rehabilitation, as it is predictive of returning to the community and of future health problems. Current research regarding post-hip fracture rehabilitation is sparse. Body weight supported treadmill training (BWSTT) is a novel approach to retrain walking abilities. BWSTT may be ideal for retraining walking after hip fracture, as it is task-specific and alleviates the demands of maintaining balance while walking skills are trained. The use of the harness may provide a sense of security for the patient, facilitating walking training. The proposed project will investigate the feasibility and tolerability of BWSTT after hip fracture, and its impact on function, mobility, quality of life and fear of falling. It is hypothesized that BWSTT 3-5 times weekly in acute hip fracture patients will improve function, mobility, quality of life and reduce fear of falling.

DETAILED DESCRIPTION:
Morbidity and mortality rates associated with hip fracture are enormous. Current literature regarding post-hip fracture rehabilitation is sparse. A recent Cochrane review suggested that the potential for enhancing the recovery of mobility in hip fracture patients with treadmill gait retraining warrants further research in this area. Body weight supported treadmill training (BWSTT) is a novel approach to retraining ambulation, and has been successfully implemented in other patient populations. BWSTT may be ideal for retraining gait after hip fracture, as it is task-specific and alleviates the demands of maintaining equilibrium while walking skills are trained. The objectives of the proposed pilot study are to evaluate the feasibility and tolerability of using BWSTT as a gait retraining strategy in individuals who have experienced a hip fracture, and to explore whether it can improve mobility, fear of falling and function. Participants' feedback will be sought regarding the BWSTT experience for use in planning future clinical trials, to be submitted to CIHR. Quantitative outcomes will be assessed at baseline, and after 4 weeks of training 3-5 times per week. Outcome measures include: the Lower Extremity Functional Scale, health-related quality of life (SF-36), Falls-Efficacy Scale and the 2-minute walk test. Based on previous research experience with the frail elderly, we anticipate that many patients will be receptive to rehabilitation in the form of BWSTT. We hypothesize that BWSTT after hip fracture will result in significant gains in ambulatory capacity, as well as improvements in quality of life and functional independence. In addition, we anticipate that BWSTT will prove to be a feasible and effective gait retraining strategy.

ELIGIBILITY:
Inclusion Criteria:

* Able to follow 2-step commands
* Stable inter-trochanteric fracture, where fixation is deemed by surgeon to be adequate, OR sub-capital fracture having undergone bipolar hemi-arthroplasty
* Able to stand and take a few steps with the help of an assistive device i.e. parallel bars, walker, or cane

Exclusion Criteria:

* Able to walk without assistive devices
* Hip, knee or ankle surgery prior to hip fracture
* Inability to understand instructions or give informed consent
* Uncontrolled cardiovascular disease or hypertension, diabetes, neuromuscular disease or other musculoskeletal disease such as rheumatoid arthritis, Uncontrolled pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora Giangregorio, PhD, Principal Investigator — University of Waterloo; Alexandra Papaioannou, MD, MSc, Principal Investigator — Hamilton Health Sciences and McMaster University
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giangregorio LM, Thabane L, Debeer J, Farrauto L, McCartney N, Adachi JD, Papaioannou A. Body weight-supported treadmill training for patients with hip fracture: a feasibility study. Arch Phys Med Rehabil. 2009 Dec;90(12):2125-30. doi: 10.1016/j.apmr.2009.06.022. PMID 19969179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients treated for a hip fracture by orthopedic surgeons and admitted to the inpatient rehabilitation floor of a teaching hospital between September 2006 and November 2007 were considered for participation. A break in recruitment was implemented from November to early January to avoid variation in physiotherapy care related to holidays.
Groups:
- Control: Usual care
Period: Baseline to Discharge
Arm/Group | BWSTT | Control
Started | 14 | 7
Completed | 12 | 5
Not Completed | 2 | 2
Not completed — not interested | 1 | 0
Not completed — MRSA | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Follow-up
Arm/Group | BWSTT | Control
Started | 12 | 5
Completed | 10 | 4
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BWSTT | Control | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.9 (7.0) | 83.7 (8.6) | 81.2 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 2 | 1 | 3
Timed up and go time [Mean (Standard Deviation); unit: seconds] — Population: Some participants could not complete performance based measures at baseline.
  seconds
    number analyzed (Participants) | 8 | 4 | 12
    (all) | 73.9 (29.1) | 45.6 (10.3) | 64.8 (27.8)
2 Minute Walk Test time [Mean (Standard Deviation); unit: metres] — Population: Some participants could not perform performance based measures at baseline
  metres
    number analyzed (Participants) | 11 | 7 | 18
    (all) | 18.7 (18.9) | 23.6 (15.3) | 20.6 (17.3)
Lower Extremity Functional Score [Mean (Standard Deviation); unit: units on a scale] — range 0-80 higher mean better functioning
  units on a scale | 16.6 (8) | 25.7 (16.5) | 19.7 (11.9)
Falls Self-efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — 0-40, higher means greater efficacy
  units on a scale | 22.4 (9.2) | 22.0 (8.2) | 22.2 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - # With > or = 60% Compliance, # Agreeing to Participate, # Returning for 3 Month Follow-up
Description: Compliance to BWSTT only,
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | BWSTT
Number analyzed (Participants) | 14
Participants
  # agreed to participate | 14
  #returned for 3 month followup | 10
  # with at least 60% compliance | 6

2. Secondary Outcome: Timed up and Go
Time Frame: discharge
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BWSTT | Control
Number analyzed (Participants) | 12 | 5
seconds | 25.2 (7.0) | 20.7 (5.0)
Statistical Analysis 1: Comparison: BWSTT vs Control; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Net) = -26.3, 95% CI 2-sided [-72.1 to 19.6]

3. Secondary Outcome: Falls Self Efficacy
Time Frame: discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BWSTT | Control
Number analyzed (Participants) | 12 | 5
units on a scale | 17.7 (6.6) | 12.8 (4.4)

4. Secondary Outcome: 2 Minute Walk Test
Time Frame: discharge
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | BWSTT | Control
Number analyzed (Participants) | 8 | 5
metres | 70.6 (17.3) | 79.4 (17.9)

5. Secondary Outcome: Lower Extremity Functional Scale
Time Frame: discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BWSTT | Control
Number analyzed (Participants) | 12 | 5
units on a scale | 35.3 (7.5) | 46.4 (7.2)
Statistical Analysis 1: Comparison: BWSTT vs Control; Test type: Superiority or Other; p = 0.40, Regression, Linear; Mean Difference (Net) = 2.8, 95% CI 2-sided [-3.6 to 9.2]

ADVERSE EVENTS:
Time Frame: inpatient stay: varies
Description: Only collected adverse events reported by participants or therapists as related to treatment as patients were already in hospital
Groups:
- Usual Care: Usual care rehabilitation
Arm/Group | BWSTT | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5
Other Adverse Events (participants affected / at risk) | 0/12 | 0/5

LIMITATIONS AND CAVEATS:
It was not possible to blind outcome assessors. We did not randomize participants because we wanted a minimum of 12 to test feasibility of intervention. Control group had a longer average length of stay, and may have received more physiotherapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No